CLINICAL TRIAL: NCT03036332
Title: Effects of Aerobic Interval Training on Clinical Biomarkers and Quality of Life in Metabolic Syndrome
Brief Title: Exercise Training and Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Rodolfo Augusto Travagin Miranda, Mr. Rodolfo Augusto Travagin Miranda, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RATMiranda1
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Metabolic Syndrome
Keywords: aerobic interval training; biomarkers
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Aerobic interval training
  Interventions: Behavioral: Aerobic interval training
- Control group (No Intervention): The participants performed only initial evaluation and at the end of the study

INTERVENTIONS:
Behavioral: Aerobic interval training — Carried out 3 times per week for 16 weeks
  Arms: intervention

SUMMARY:
The present study aimed to determine the effects of 16 weeks of aerobic interval training on quality of life and a set of clinical biomarkers.

DETAILED DESCRIPTION:
Besides the traditional metabolic syndrome risk factors (dyslipidemia, raised blood pressure, central obesity and dysglycemia) subclinical disorders related to chronic inflammation and cell damage have been reported on metabolic syndrome. Therefore, regarding the systemic feature of metabolic syndrome, we investigated an new approach of aerobic interval training on several clinical biomarkers widely used. Such training used differs from current aerobic protocols in order to attenuate metabolic and musculoskeletal overload on untrained and unhealthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Having metabolic syndrome according to international diabetes foundations definition (IDF).
* Age between 35 - 60 years and untrained subjects.

Exclusion Criteria:

* Musculotendinous or osteoarticular injuries in the lower limbs and/or spine
* Chronic pulmonary diseases
* Neurological disorders
* Kidney failure
* High-risk cardiovascular diseases (Unstable angina pectoris, Uncompensated heart failure, complex ventricular arrhythmias or myocardial infarction during the last month).

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-12-10 (Actual); Study Completion 2016-12-10 (Actual)

PRIMARY OUTCOMES:
Pro-inflammatory marker | 16 weeks
  Serum levels of C-reactive protein

SECONDARY OUTCOMES:
Quality of life | 16 weeks
  The Medical Outcomes Study-Short Form 36 (SF-36)
A set of clinical biomarkers | 16 weeks
  Serum levels lof Homocysteine; Creatinine, Creatine kinase (ck); creatine kinase MB (ck-mb); Troponin t; aspartate aminotransferase; alanine aminotransferase; and complete blood count.

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo AT Miranda, Me, Principal Investigator — Universidade Estadual Paulista Júlio de Mesquita

IPD SHARING:
Plan to Share IPD: No